CLINICAL TRIAL: NCT07261423
Title: Pollution Intervention to Impact Kids Asthma Study
Acronym: PIKAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Franziska Rosser, MD MPH, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY25060085; R01ES036965 (NIH)
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Childhood Asthma; Asthma Control; Asthma Exacerbation; Air Pollution, Risk Reduction Behaviors
Keywords: childhood asthma; air quality index; AQI
MeSH Terms: conditions — Risk Reduction Behavior | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Unblinded, randomized controlled parallel trial, stratified by age group (8-12 year, 13-17 year).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Standard outdoor air pollution education + asthma action plan) (Active Comparator): Control
  Interventions: Behavioral: Education and plan
- EPA-AQI (Education+ plan + EPA-AQI) (Experimental): EPA-AQI
  Interventions: Behavioral: EPA-AQI; Behavioral: Education and plan
- Commercial-AQI (Education+ plan + commercial-AQI) (Experimental): Commercial-AQI
  Interventions: Behavioral: Commerical-AQI; Behavioral: Education and plan

INTERVENTIONS:
Behavioral: EPA-AQI — The EPA-AQI group will receive standardized outdoor air pollution education, standardized AQI education, instructions for AQI usage, and an asthma action plan containing information specific for the EPA-AQI, and will demonstrate the ability to navigate to the EPA-AQI via smartphone app or website.
  Arms: EPA-AQI (Education+ plan + EPA-AQI)
Behavioral: Commerical-AQI — The commercial-AQI group will receive standardized AQI education, instructions for commercial-AQI usage, and an asthma action plan containing information specific for the commercial-AQI, and will demonstrate the ability to navigate to the commercial-AQI via smartphone or website.
  Arms: Commercial-AQI (Education+ plan + commercial-AQI)
Behavioral: Education and plan — Standardized outdoor air pollution education and standard asthma action plan

SUMMARY:
The goal of this clinical trial is to learn if adding Air Quality Index (AQI) information to asthma action plans works to improve asthma outcomes in children. It will also learn about children with asthma who report being more sensitive to outdoor air pollution. The main questions it aims to answer are:

* Does adding either information about the EPA-AQI or commercial AQI improve asthma outcomes over time?
* Are there changes in nasal gene expression in children with asthma who report they are more sensitive to outdoor air pollution?

Researchers will compare EPA-AQI and the commercial-AQI groups to a control group to either AQI works to improve asthma.

Participants will:

* Receive standardized outdoor air pollution education and an asthma action plan
* Provide nose and blood specimens
* Have visits every 4 weeks for 48 weeks, 10 will be conducted by telephone calls and 3 visits will be in person.

ELIGIBILITY:
Inclusion Criteria:

* A healthcare provider diagnosis of persistent asthma (Steps 2-5 as defined by US guidelines) or intermittent asthma (Step 1) + at least one severe asthma exacerbation (defined by American Thoracic Society (ATS)/European Respiratory Society (ERS) criteria as requiring at least 3 days of systemic steroids or an Emergency Department/Urgent Care visit requiring systemic steroids) in the prior 12 months
* Home access to a smartphone or internet
* Primary residence in Allegheny County, PA
* One participant per household
* Age 8 -17 years
* Healthcare provider evaluation for asthma in the prior year

Exclusion Criteria:

* Diagnosis of other active chronic respiratory diseases (e.g., cystic fibrosis, bronchopulmonary dysplasia, etc.)
* Neuromuscular disorder
* Chronic disorder limiting independent ambulation (e.g., spastic quadriplegia, etc.)
* Cyanotic heart disease
* Plans to relocate from Allegheny County, PA in the next year (12 months)
* Use of intranasal or oral/intramuscular/intravenous corticosteroids 4 weeks prior to randomization
* Current participation in another asthma intervention trial

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 351 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Change in asthma control scores, over-time, between groups | Baseline through 48 weeks, measured at 4 week intervals
  Asthma control will be measured via the validated Asthma Control Test (ACT) and Childhood-ACT (CACT). Asthma control will be evaluated at all study visits (Visits 1-13), every 4 weeks. The ACT will be used for children aged 12 -17 years, the CACT will be used for children aged 8-11 years. The ACT is a 5 question instrument with scores from 5-25, with higher scores generally indicating better control. The CACT is a 7 question instrument with scores from 0-27, with higher scores generally indicating better control. For both ACT and CACT, scores of 19 or less are concerning for poor asthma control and both measure control in the past 4 weeks.

SECONDARY OUTCOMES:
Change in Pediatric Asthma Quality of Life (PAQLQ) score over-time between groups | Baseline through 48 weeks, measured at Visit 1 (time=0), Visit 7 (time=24 weeks), and Visit 13 (time=48 weeks).
  Asthma quality of life will be measured using the validated Pediatric Asthma Quality of Life Questionnaire (PAQLQ) and administered by research coordinators at all in-person visits: randomization (Visit 1), Visit 7 (24 weeks), and exit (Visit 13). The PAQLQ ranges from 1 to 7, with higher scores indicating higher quality of life.
Severe asthma exacerbations, having at least one, over-time between groups | Baseline through 48 weeks, measured at 4 week intervals
  Self-reported severe asthma exacerbations (SAE) will be measured every 4 weeks via questionnaire, administered at all study visits (Visits 1- 13). SAE are defined by American Thoracic Society criteria and include increased asthma symptoms requiring at least 3 days of systemic steroids OR increased asthma symptoms for which Emergency Department or Urgent Care evaluation was sought and for which systemic steroids were administered/prescribed). SAE will be categorized as yes or no for a study visit.

OTHER OUTCOMES:
Differential nasal gene expression in children with asthma reporting increased susceptibility to outdoor air pollution | Baseline through 48 weeks, measured at 4 week intervals
  A component of our EPA-AQI and commercial-AQI intervention is to encourage participants to learn their own personal susceptibility to outdoor air pollution. We will assess if participants report symptoms to specific AQI categories at all visits via questionnaire (yes, no). Questionnaires are administered every 4 weeks at all study visits (Visits 1-13). Transcriptome-wide differential gene expression (obtained at baseline visit) will be compared between children who report low susceptibility to specific AQI category versus those who do not, with susceptibility being defined by reported susceptibility during the 48 week study, measured every 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Franziska Rosser, MD MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Select de-identified data will be made available after study completion and as per Data Management and Sharing Plan.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified data generated from this project will be made available no later than the time of publication or the end of the funding period, whichever comes first.
Access Criteria: Raw data and identifiable data will not be shared except where institutional agreements, certifications, and informed consent allows. De-identified data will be available by controlled access only within data repositories.